CLINICAL TRIAL: NCT01320371
Title: Clinical Outcomes and Cost Analysis of Standard Versus Barbed Sutures for Closure in Primary Total Knee Arthroplasty: A Single Blinded Multicenter Prospective Randomized Trial.
Brief Title: Analysis of Standard Versus Barbed Sutures in Primary Total Knee Arthroplasty.
Status: Completed | Type: Observational
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Christopher Peters, M.D., University of Utah
Other Study IDs: 44725
Record Dates: First submitted 2011-03-18; First posted 2011-03-22 (Estimated); Last update posted 2014-02-04 (Estimated); Status verified 2014-02

CONDITIONS: Arthropathy of Knee
Keywords: barbed sutures; knotted sutures; total knee arthroplasty; knee surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Barbed sutures: Barbed sutures are self-anchoring, requiring no knots for wound closure.
- Knotted sutures: Knotted sutures used for traditional surgical closures.

SUMMARY:
The purpose of this prospective study is determine if barbed sutures are more efficient, have comparable complication rates, clinical outcomes, and cosmesis outcomes versus traditional knotted sutures when used in the closure of primary total knee arthroplasty (TKA).

Barbed suture has been associated with improved closure efficiency and safety in TKA in prior studies. The investigators performed a multicenter randomized controlled trial to determine the efficiency and safety of this technology in TKA. The investigators prospectively randomized 411 patients undergoing primary TKA to either barbed running (n=191) or knotted interrupted suture closure (n=203). Closure time was measured intraoperatively. Cost analysis was based on suture and operating room time costs.

DETAILED DESCRIPTION:
Total knee arthroplasty (TKA) rates have consistently risen in recent years, and demand is expected to increase by over 600% in the next 20 years. Decreasing reimbursement and available resources make tangible advances in surgical efficiency and outcomes essential in meeting current and future demand. Closure time may be one of the best targets in the push to reduce operative time and cost while increasing operative productivity. Optimizing lengthy, multilayered wound closures in TKA is a promising means for improving both efficiency and outcomes by potentially decreasing wound closure time, reducing postoperative wound complications, and improving cosmetic outcomes.

Running knotless suture technique utilizing barbed suture technology has recently been shown to reduce wound closure time in both total hip and knee arthroplasty in a small, prospective, randomized clinical trial. Barbed suture technology has also facilitated rapid closure and soft-tissue repair in plastic-surgery literature. Very few studies have reported on the use of barbed suture technology for multilayered closure in orthopedics. As a pilot study, the investigators performed a retrospective analysis of consecutive cohorts before and after changing to barbed suture. The investigators believed that our published slight improvement in efficiency and cost savings of a barbed suture closure was underestimated due to the retrospective nature of our pilot study and the investigators therefore elected to proceed forward with a prospective randomized trial. Additionally, in the investigators pilot study we found a potential trend toward lower wound complications with the barbed suture and we wanted to see if this would be borne out in a prospective randomized trial.

The investigators hypothesized that a prospective study would show that barbed sutures would be more efficient, have comparable complication rates, clinical outcomes, and cosmesis outcomes versus traditional knotted sutures when used in the closure of primary TKA. Specifically, the investigators hypotheses were as follows: multilayered closure in TKA with barbed suture would be associated with (1) shorter closure times; (2) lower cost; (3) similar closure related perioperative complication rates; and (4) similar Knee Society, cosmesis, and patient satisfaction scores when compared to standard knotted suture closure.

ELIGIBILITY:
Inclusion Criteria:

* Patients greater than 18 years of age
* Undergoing primary total knee arthroplasty
* English speaking

Exclusion Criteria:

* Patients less than 18 years of age
* Prior open knee surgery in close proximity (<2cm) to the proposed incision for the primary total knee arthroplasty (prior arthroscopic surgery does not exclude a patient from the study)
* Wound or Scar in close proximity (<2cm) to the proposed incision for the primary total knee arthroplasty

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study and control groups will be made up of consecutive patients undergoing a median parapatellar approach primary total knee arthroplasty at the University of Utah Hospital and Clinics. The control group will undergo two-layer closure utilizing a standard interrupted, knotted suture technique. The closures will be performed by 2 members of the team (attending surgeon, resident, fellow, or PA) in ALL closures so as to limit the possible confounder of closure time variation due to different numbers of people closing the incision. This will specifically consist of arthrotomy closure using interrupted #1 Ethibond™ in figure of eight fashion and sudermal closure using 2-0 Monocryl™ in interrupted buried fashion.
Sampling Method: Non-Probability Sample
Enrollment: 363 (Actual)
Dates: Start 2011-01; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Intraoperative closure time in total knee arthroplasty. | 6 weeks

SECONDARY OUTCOMES:
Cost analysis in terms of operative time and material costs of closure in total knee arthroplasty. | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Peters, MD, Principal Investigator — University of Utah hopsital; Jeremy Gililland, MD, Principal Investigator — University of Utah Orthopaedics Resident
Locations (4):
- United States (4):
  - Duke University Health System, Durham, North Carolina
  - Joint Implant Surgeons Inc,, New Albany, Ohio
  - Scott and White HealthCare, Temple, Texas
  - University of Utah Orthopedics Center, Salt Lake City, Utah